CLINICAL TRIAL: NCT03935295
Title: Dysport ® (abobotulinumtoxinA) as an Adjunctive Treatment to Bracing in the Management of Adolescent Idiopathic Scoliosis
Brief Title: Dysport ® as an Adjunctive Treatment to Bracing in the Management of Adolescent Idiopathic Scoliosis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00110399
Record Dates: First submitted 2019-04-30; First posted 2019-05-02 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: AIS; adolescent idiopathic scoliosis
MeSH Terms: interventions — abobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Botulinum Toxin (Experimental): The investigators plan to administer approximately 1000 U Dysport ® in the concave-sided paraspinal musculature of the major curve, based on an estimated total dose of 1000 U, the maximum allowable dose. The total dose per treatment session will not exceed 15 units/kilogram or 1000 units, whichever is lower. If two curves are equivalent within 3˚, both will be treated, however, the dosing (described above) will be divided equally across both curves.
  There will be two cycles of injections. Patients will be treated at time 0 (baseline) and 4 months.
  Interventions: Drug: AbobotulinumtoxinA; Device: Custom Thoracolumbosacral Orthosis
- Placebo (Placebo Comparator): Control patients will receive an injection of placebo specifically prepared as a control for this study. The same volumes as indicated in the "experimental" arm description will be injected.
  These will be administered during two cycles of injections. Patients will be treated at time 0 (baseline) and 4 months.
  Interventions: Drug: Placebos; Device: Custom Thoracolumbosacral Orthosis

INTERVENTIONS:
Drug: AbobotulinumtoxinA — Paraspinal abobotulinumtoxinA injections (compared to placebo)
  Other Names: Dysport, Ipsen
  Arms: Botulinum Toxin
Drug: Placebos — Placebo prepared by Ipsen for use as control
  Arms: Placebo
Device: Custom Thoracolumbosacral Orthosis — Non-operative external bracing for scoliosis curves

SUMMARY:
This study evaluates the combined effect of botulinum toxin A (administered as Dysport® (Ipsen Pharmaceuticals)) and bracing in children with adolescent idiopathic scoliosis. Two thirds of patients will be treated with Dysport® and bracing, while the remaining patients will be treated with placebo and bracing.

DETAILED DESCRIPTION:
Adolescent idiopathic scoliosis (AIS) is lateral curvature of the spine with an unknown cause in children 10-16 years old. Without treatment, skeletally immature children with idiopathic curves of 20°-40° risk curve progression. Treatment of these patients is focused on either observation or bracing. Although bracing has been shown to be more effective than observation, success is contingent on patient adherence and has the potential for further optimization with adjunct therapies.

Little research is available concerning adjunct therapies that may be used during bracing of AIS patients. One therapy in particular, abobotulinumtoxinA (BTX) injection, has been poorly studied. Injection of BTX into the paraspinal musculature of the concave aspect of the major curve may result in a more malleable curve and thus optimize brace treatment. If BTX injections are found to improve outcomes in this way, a new standard of nonoperative care could be established for AIS patients, potentially reducing the number of patients who undergo surgery.

The aim of this study is to assess whether BTX injections (administered as Dysport® (Ipsen Pharmaceuticals)) in the paraspinal musculature at the site of the major scoliotic curve decrease curve progression in skeletally immature AIS patients who are concurrently treated with bracing. Dysport® will be evaluated primarily as an adjunct treatment to bracing.

Hypotheses

1. Dysport® injections into the concave-side paraspinal muscles will decrease the rate of curve progression, with a lower rate of curve progression in patients treated with both Dysport® injections and bracing compared with those treated with only bracing.
2. Quantitative physical and mental health scores will improve to a greater extent in patients treated with Dysport® and bracing compared with patients treated with only bracing.

ELIGIBILITY:
Inclusion criteria:

* Clinically determined idiopathic nature of scoliosis
* Age 10-16 years
* Risser stage 0,1,or 2
* major curve of 20°-40°
* curve apex caudal to T7 vertebra
* ability to adhere to bracing protocol
* Botulinum toxin naïve or previously treated greater than 6 months prior to study entry

Exclusion criteria:

* Diagnosis of congenital scoliosis, neuromuscular scoliosis, or other "reason" for scoliosis - Previous surgery at any segment of the spine
* Current need for surgery at any level of the spine
* Treatment with any drug known to interfere with neuromuscular function
* Any other medical condition, laboratory or diagnostic procedure finding that might preclude administration of BTX
* Ongoing infection at the injection sites
* Diagnosis as either resistant or sensitive to botulinum toxin treatment of any type or to any components of the BTX formulation
* Cow milk protein allergy

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2020-09-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in scoliotic curve as assessed by the Major Curve Cobb Angle | Assessed at baseline (time 0), 6 weeks, 4 months, 4 months + 6 weeks, 8 months
  Change in scoliotic curve will be assessed using by the Major Curve Cobb Angle with measurement of standing scoliosis radiographs. Cobb angle refers to a radiographic measurement of side to side spinal curvature, measured in angle degrees.

SECONDARY OUTCOMES:
Change in Patient Reported Outcomes | Assessed at baseline (time 0), 6 weeks, 4 months, 4 months + 6 weeks, 8 months
  This will be assessed by Scoliosis Research Society (SRS) 22 Survey; The SRS-22 questionnaire is a validated measure used to assesses quality of life in patients with idiopathic scoliosis. It consists of five domains that assess: function, pain, mental health, self-image, and satisfaction with treatment. Higher scores indicate increased satisfaction. Each of the 22 questions are scored on a scale of 1 to 5.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sponseller, MD, MBA, Principal Investigator — Johns Hopkins Hospital Department of Orthopaedic Surgery; Varun Puvanesarajah, MD, Principal Investigator — Johns Hopkins Hospital Department of Orthopaedic Surgery
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hresko MT. Clinical practice. Idiopathic scoliosis in adolescents. N Engl J Med. 2013 Feb 28;368(9):834-41. doi: 10.1056/NEJMcp1209063. No abstract available. PMID 23445094
- [Background] Asher MA, Burton DC. Adolescent idiopathic scoliosis: natural history and long term treatment effects. Scoliosis. 2006 Mar 31;1(1):2. doi: 10.1186/1748-7161-1-2. PMID 16759428
- [Background] Weinstein SL. Idiopathic scoliosis. Natural history. Spine (Phila Pa 1976). 1986 Oct;11(8):780-3. doi: 10.1097/00007632-198610000-00006. PMID 3810292
- [Background] Weinstein SL, Dolan LA. The Evidence Base for the Prognosis and Treatment of Adolescent Idiopathic Scoliosis: The 2015 Orthopaedic Research and Education Foundation Clinical Research Award. J Bone Joint Surg Am. 2015 Nov 18;97(22):1899-903. doi: 10.2106/JBJS.O.00330. No abstract available. PMID 26582623
- [Background] Weinstein SL, Dolan LA, Wright JG, Dobbs MB. Effects of bracing in adolescents with idiopathic scoliosis. N Engl J Med. 2013 Oct 17;369(16):1512-21. doi: 10.1056/NEJMoa1307337. Epub 2013 Sep 19. PMID 24047455
- [Background] Nuzzo RM, Walsh S, Boucherit T, Massood S. Counterparalysis for treatment of paralytic scoliosis with botulinum toxin type A. Am J Orthop (Belle Mead NJ). 1997 Mar;26(3):201-7. PMID 9240788
- [Background] Wong C, Gosvig K, Sonne-Holm S. The role of the paravertebral muscles in adolescent idiopathic scoliosis evaluated by temporary paralysis. Scoliosis Spinal Disord. 2017 Oct 10;12:33. doi: 10.1186/s13013-017-0138-7. eCollection 2017. PMID 29046898
- [Background] Kouwenhoven JW, Castelein RM. The pathogenesis of adolescent idiopathic scoliosis: review of the literature. Spine (Phila Pa 1976). 2008 Dec 15;33(26):2898-908. doi: 10.1097/BRS.0b013e3181891751. PMID 19092622
- [Background] Wong C. Mechanism of right thoracic adolescent idiopathic scoliosis at risk for progression; a unifying pathway of development by normal growth and imbalance. Scoliosis. 2015 Jan 27;10:2. doi: 10.1186/s13013-015-0030-2. eCollection 2015. PMID 25657814
- [Background] RIDDLE HF, ROAF R. Muscle imbalance in the causation of scoliosis. Lancet. 1955 Jun 18;268(6877):1245-7. doi: 10.1016/s0140-6736(55)91020-5. No abstract available. PMID 14382561
- [Background] Fidler MW, Jowett RL. Muscle imbalance in the aetiology of scoliosis. J Bone Joint Surg Br. 1976 May;58(2):200-1. doi: 10.1302/0301-620X.58B2.932082.
- [Background] Asher M, Min Lai S, Burton D, Manna B. The reliability and concurrent validity of the scoliosis research society-22 patient questionnaire for idiopathic scoliosis. Spine (Phila Pa 1976). 2003 Jan 1;28(1):63-9. doi: 10.1097/00007632-200301010-00015. PMID 12544958
- [Background] Cheung KM, Cheng EY, Chan SC, Yeung KW, Luk KD. Outcome assessment of bracing in adolescent idiopathic scoliosis by the use of the SRS-22 questionnaire. Int Orthop. 2007 Aug;31(4):507-11. doi: 10.1007/s00264-006-0209-5. Epub 2006 Aug 1. PMID 16896864
- [Background] Schwieger T, Campo S, Weinstein SL, Dolan LA, Ashida S, Steuber KR. Body Image and Quality-of-Life in Untreated Versus Brace-Treated Females With Adolescent Idiopathic Scoliosis. Spine (Phila Pa 1976). 2016 Feb;41(4):311-9. doi: 10.1097/BRS.0000000000001210. PMID 26555827
- [Background] Wong C, Pedersen SA, Kristensen BB, Gosvig K, Sonne-Holm S. The Effect of Botulinum Toxin A Injections in the Spine Muscles for Cerebral Palsy Scoliosis, Examined in a Prospective, Randomized Triple-blinded Study. Spine (Phila Pa 1976). 2015 Dec;40(23):E1205-11. doi: 10.1097/BRS.0000000000001049. PMID 26165216